CLINICAL TRIAL: NCT05908422
Title: Alvision™ Interventional Cardiology Diagnostic Catheter Use for Routine Diagnostic Procedures in Angiographic Applications: Evaluation of Safety and Performance in Everyday Clinical Practice. The Alvision™ Interventional Cardiology Diagnostic Catheter Post Market Clinical Follow-up (PMCF) Study.
Brief Title: The Alvision™ Interventional Cardiology Diagnostic Catheter Post Market Clinical Follow-up (PMCF) Study.
Status: Completed | Type: Observational
Sponsor: Alvimedica (Industry)
Responsible Party: Sponsor
Other Study IDs: C42102
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Coronary Disease; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Alvision™ Interventional Cardiology Diagnostic Catheter — The Alvision™ Interventional Cardiology Diagnostic Catheter is a single use only, thin, flexible single lumen tube, with a proximal hub, sterilized with ethylene oxide (EO) gas, non-pyrogenic. The product is defined as a catheter to inject a contrast medium into selected blood vessels.

SUMMARY:
The objective of this prospective observational study is to collect clinical data on the medical device Alvision™ Interventional Cardiology Diagnostic Catheter in an unselected population in the current clinical practice

DETAILED DESCRIPTION:
Within the scope of this observational medical device trial, brand/model of the catheter that will be used during the PCI will be decided by the physician and decision of the physician won't be interfered. PCI will be performed according to the standard clinical procedures. Data of the patients to whom Alvision™ Interventional Cardiology Diagnostic Catheter is applied will be gathered for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Turkish citizen,
* ≥18 years of age,
* Has indication for a diagnostic coronarography according to Alvision™ Instruction for use,
* Has signed and dated the informed consent.

Exclusion Criteria:

* Having a known allergic reaction to any of the composition of Alvision™ Interventional Cardiology Diagnostic Catheter.
* Has synthetic vascular grafts through which the Alvision™ Interventional Cardiology Diagnostic Catheter should pass
* Participating in another medical device or pharmaceutical clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of all patients in which the Alvision™ Interventional Cardiology Diagnostic Catheter is used who meet the study inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Ratio of the successful delivery of radio-opaque media to selected sites in the coronary vascular system. | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
Major adverse cardiovascular events (MACEs) and stroke associated with the use of diagnostic catheters until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure, whichever happens first: | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
  * Thrombus formation/emboli
  * Arterial wall damage
  * Myocardial infarction
  * Plaque dislodgement
  * Cardiac arrhythmia
  * Death
  * Stroke

SECONDARY OUTCOMES:
Ratio of the successfully insertion catheter | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
Capacity of providing the doctor with a safe and effective tool to perform angiographies | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
  * Ratio of damage on vessels (%)
  * Ratio of cardiogenic shock (%)
  * Ratio of the straight course of the catheter through the vessels (%)
Duration of the various stages the procedure (before the procedure, during and after the procedure) and a qualitative and quantitative assessment of angiographic quality | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
  * Trackability (%)
  * Torquability (%) ,
  * Slippage (%) ,
Ratio of the total volume of radio-opaque media delivered to the planned amount of using volume | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
Determination of the relation between catheter size, and patients' height. | until discharge from hospital or 24 hours after PCI (Percutaneous Coronary Intervention) procedure
  catheter size (cm) patients' height (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Alvimedica, Istanbul, Turkey (Türkiye)